CLINICAL TRIAL: NCT06039358
Title: Influence of 6mg/kg of Caffeine Supplementation on the Technical Execution of General Movement Patterns Performed by Healthy Subjects, With and Without Neuromuscular Fatigue: a Randomized, Double-blind, Placebo-controlled, Crossover Trial
Brief Title: Effects of Caffeine Ingestion on the Biomechanics of Healthy Young Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: Generalitat de Catalunya (Unknown); European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CAFBIOM001
Record Dates: First submitted 2023-09-01; First posted 2023-09-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Caffeine; Biomechanics; Fatigue; Injuries; Physical Activity
Keywords: Ergogenic aids; Kinematics; Kinetics; Neuromuscular fatigue; Acute and chronic injuries; Jump; Squat; Running
MeSH Terms: conditions — Fatigue; Wounds and Injuries; Motor Activity | interventions — Caffeine; Cellulose

STUDY DESIGN:
Intervention Model Description: The assessed sessions, which will be identical, will be the control, the caffeine, and the placebo ones. The last two sessions mentioned will be performed in a randomized order.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The placebo and the caffeine ingestion protocols will be identical in format and presentation. To minimize any influence of the flavor or the look of the ingested substance, both conditions will imply the consumption of opaque capsules (ingested with water) in which there will be 6mg/kg of caffeine or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - caffeine - placebo. (Experimental): The order of the assessed sessions will be first the control one, then the caffeine one, and then the placebo one.
  Interventions: Dietary Supplement: Caffeine.; Drug: Cellulose.
- Control - placebo - caffeine. (Experimental): The order of the assessed sessions will be first the control one, then the placebo one, and then the caffeine one.
  Interventions: Dietary Supplement: Caffeine.; Drug: Cellulose.

INTERVENTIONS:
Dietary Supplement: Caffeine. — Ingestion of opaque capsules with a total dose of 6mg/kg of caffeine, 60 minutes before the beginning of the assessed exercises. A crossover with the other intervention will be done in the next/previous session (depending on the arm).
Drug: Cellulose. — Ingestion of opaque capsules with cellulose, 60 minutes before the beginning of the assessed exercises. A crossover with the other intervention will be done in the next/previous session (depending on the arm).
  Other Names: Placebo.

SUMMARY:
Caffeine is one of the few supplements that have enough scientific evidence to state that can notably improve performance, as different remarkable organizations in the sports nutrition context have classified it as an ergogenic aid with strong evidence regarding its efficacy and that is apparently safe. The beneficial effect of this substance on physical and cognitive performance has been identified in aerobic and anaerobic efforts, including aerobic and muscular endurance, power, or strength.

However, it seems that the benefits of caffeine are usually measured only by its effect on performance, while a comprehensive analysis of its impact on other aspects of the movement technique of the exercise is not considered. Therefore, although caffeine generates better performance, a null or negative effect may occur on technique execution. As such, some consequences might arise (e.g., an increase in injury risk or a decrease in energy efficiency).

The objective of this randomized controlled trial is to assess the influence of caffeine on certain biomechanical parameters of the technique of physical exercises in circumstances without fatigue and under neuromuscular fatigue. The study hypothesis is that caffeine generates modifications in the technical execution of certain movements in fatigued and unfatigued circumstances due to its physiological effects, which may be beneficial for performance and injury prevention.

The participants will have to attend 5 sessions (enrollment, familiarization, control, placebo, and caffeine), at least 7 days apart. In the last 3 sessions, different measurements will be done to their technique while jumping, squatting, and running, without fatigue and with it. Other data will be collected throughout the study to contextualize and analyze in more detail the obtained information.

DETAILED DESCRIPTION:
A detailed description of the study can be found in the protocol uploaded with this registry entry.

ELIGIBILITY:
Inclusion Criteria:

* An uninterrupted training time of at least 1 year in the subjects' regular exercise modality (either the person is still training or interrupted the training period during the last year, and with no more than 4 months of detraining).
* A good exercise technique of the assessed movement patterns (running, squatting, and jumping).

Exclusion Criteria:

* Not being 18-30 years old.
* Having any relevant medical condition.
* Pregnancy.
* Smoking.
* Regular medication consumption / Medication consumption the days before the sessions during the study.
* Other supplementation regular consumption / Other supplementation consumption during the study (excluding sports foods, provided that their goal and nutrients have the objective of substituting the ingestion of regular food (e.g., isotonic drinks, carbohydrates gels, protein powder...), without adding other components that may act as ergogenic substances).
* Habitual caffeine consumption of >25mg/day-0,99mg/kg/day.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Knee flexion angle at the midstance while running. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the knee flexion angle (in degrees). The measurement will be done before and after a fatiguing protocol. Assessed using kinematic instruments.
Ankle dorsiflexion angle at the midstance while running. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the ankle dorsiflexion angle (in degrees). The measurement will be done before and after a fatiguing protocol. Assessed using kinematic instruments.
Step rate while running. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the step rate (in steps/minute). The measurement will be done before and after a fatiguing protocol. Assessed using kinematic instruments.
Contact time while running. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the time the foot is in contact with the ground (in seconds). The measurement will be done before and after a fatiguing protocol. Assessed using kinematic instruments.
Stride length while running. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the distance between two successive placements of the same foot (in meters). The measurement will be done before and after a fatiguing protocol. Assessed using kinematic instruments.
Flight time while running. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the time the foot is not in contact with the ground (in seconds). The measurement will be done before and after a fatiguing protocol. Assessed using kinematic instruments.
Running performance modification. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the time (in seconds) required to complete a specific distance running on a treadmill. The measurement will be done before and after a fatiguing protocol. Assessed using a stopwatch.
Hip angle while squatting, at the initial position, bottom position, and final position, and the eccentric and the concentric range of movement. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the hip angle (in degrees). The measurement will be done before and after a fatiguing protocol. Assessed using kinematic instruments.
Knee angle while squatting, at the initial position, bottom position, and final position, and the eccentric and the concentric range of movement. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the knee angle (in degrees). The measurement will be done before and after a fatiguing protocol. Assessed using kinematic instruments.
Ankle angle while squatting, at the initial position, bottom position, and final position, and the eccentric and the concentric range of movement. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the ankle angle (in degrees). The measurement will be done before and after a fatiguing protocol. Assessed using kinematic instruments.
Execution time while squatting, for the eccentric and the concentric phases of the movement. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the execution time to perform the eccentric and the concentric phases of the squat (in seconds). The measurement will be done before and after a fatiguing protocol. Assessed using a linear position transducer.
Peak vertical force while squatting, for the eccentric and the concentric phases of the movement. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the peak vertical force (in Newtons). The measurement will be done before and after a fatiguing protocol. Assessed using a linear position transducer.
Rate of force development while squatting, for the eccentric and the concentric phases of the movement. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the rate of force development (in Newtons/seconds). The measurement will be done before and after a fatiguing protocol. Assessed using a linear position transducer.
Squatting performance modification. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the mean propulsive bar velocity (in meters/seconds) for a specific weight lifted in barbell back squats. The measurement will be done before and after a fatiguing protocol. Assessed using a linear position transducer.
Contralateral pelvic drop angle while jumping, at the initial contact of the landing phase. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the contralateral pelvic drop angle (in degrees). The measurement will be done before and after a fatiguing protocol. Assessed using kinematic instruments.
Knee valgus while jumping, at the initial contact and the deepest landing position of the landing phase, and the range of movement between these two moments. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the knee valgus angle (in degrees). The measurement will be done before and after a fatiguing protocol. Assessed using kinematic instruments.
Unweighting phase duration while jumping (jumping phase). | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the unweighting phase duration (in seconds). The measurement will be done before and after a fatiguing protocol. Assessed using force plates.
Braking phase duration while jumping (jumping phase). | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the braking phase duration (in seconds). The measurement will be done before and after a fatiguing protocol. Assessed using force plates.
Propulsive phase duration while jumping (jumping phase). | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the propulsive phase duration (in seconds). The measurement will be done before and after a fatiguing protocol. Assessed using force plates.
Relative peak power output while jumping (jumping phase). | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the relative peak power output (in Watts/kg). The measurement will be done before and after a fatiguing protocol. Assessed using force plates.
Jumping performance modification. | During the control, placebo, and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the height (in meters) of countermovement jumps. The measurement will be done before and after a fatiguing protocol. Assessed using force plates.

SECONDARY OUTCOMES:
Supplementation identification. | During the placebo and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the participants' perception regarding the ingested substance. They will have to complete a questionnaire immediately before (1 hour post-supplementation) and after the assessed exercises, indicating what substance they believe that they have consumed, with the options "caffeine", "placebo", or "I don't know", as well as the reason why they have chosen that answer.
Side effects. | During the day after the placebo and caffeine sessions (at least 7 days between them). The length of each session will be approximately 3 hours.
  Assessment of the participant's side effects related to caffeine consumption. In the morning of the day after the sessions, they will be requested to complete a questionnaire comprised of 8 questions with a yes/no answer, to evaluate the side effects of caffeine consumption during the hours after the sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Arnau Baena Riera, MSc., Principal Investigator — Sport, Exercise, and Human Movement (SEaHM), University of Vic - Central University of Catalonia.
Locations (1):
- University of Vic - Central University of Catalonia., Vic, Barcelona., Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT06039358/Prot_000.pdf